CLINICAL TRIAL: NCT01966601
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Ranging Study to Explore the Efficacy of TRV027 in Patients Hospitalized for Acute Decompensated Heart Failure
Brief Title: A Study to Explore the Efficacy of TRV027 in Patients Hospitalized for Acute Decompensated Heart Failure
Acronym: BLAST-AHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP027.2002
Record Dates: First submitted 2013-09-02; First posted 2013-10-21 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Sar-Arg-Val-Tyr-Ile-His-Pro-Ala-OH

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TRV027 dose #1 (Experimental): TRV027 dose #1 via continuous IV infusion
  Interventions: Drug: TRV027 Dose #1
- TRV027 dose #2 (Experimental): TRV027 dose #2 via continuous IV infusion
  Interventions: Drug: TRV027 Dose #2
- TRV027 dose #3 (Experimental): TRV027 dose #3 via continuous IV infusion
  Interventions: Drug: TRV027 Dose #3
- Placebo (Placebo Comparator): Placebo via continuous IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRV027 Dose #1 — TRV027 continuous intravenous infusion Dose #1
  Other Names: Formerly known as TRV120027
  Arms: TRV027 dose #1
Drug: TRV027 Dose #2 — TRV027 continuous intravenous infusion Dose #2
  Other Names: Formerly known as TRV120027
  Arms: TRV027 dose #2
Drug: TRV027 Dose #3 — TRV027 continuous intravenous infusion Dose #3
  Other Names: Formerly known as TRV120027
  Arms: TRV027 dose #3
Drug: Placebo — Placebo continuous intravenous infusion
  Arms: Placebo

SUMMARY:
To evaluate the overall safety and efficacy of TRV027 when administered in addition to standard of care (SOC) on mortality, morbidity, dyspnea, and length of stay in patients hospitalized with Acute Decompensated Heart Failure (ADHF).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥21 years and ≤ 85 years 1a.Women of non-child-bearing potential
2. Able to provide written informed consent
3. Pre-existing diagnosis of heart failure and at least 30 days treatment with daily oral loop diuretics
4. Systolic blood pressure ≥105 mmHg and ≤ 160 mmHg within 30 minutes of randomization
5. Ventricular rate ≤125 bpm. Patients with rate-controlled persistent or permanent atrial fibrillation (aFib) at screening are permitted.
6. Presence of ADHF defined by:

   * BNP > 400 pg/mL or NT-proBNP > 1600 pg/mL

     * For patients with BMI >30 kg/m2: BNP > 200 pg/mL or NT-proBNP > 800 pg/mL
     * For patients with rate-controlled persistent or permanent aFib: BNP > 600 pg/mL or NT-proBNP > 2400 pg/mL
     * Congestion on chest radiograph (CXR)

   AND at least two (2) of the following:
   * Rales by chest auscultation
   * Edema ≥ +1 on a 0-3 + scale, indicating indentation of skin with mild digital pressure that requires 10 or more seconds to resolve in any dependent area including extremities or sacral region.
   * Elevated jugular venous pressure (≥8 cm H2O)
7. Receipt of a IV loop diuretic at a minimum dose 40 mg furosemide (or equivalent loop diuretic) for the treatment of dyspnea due to ADHF at least 1 hour prior to anticipated randomization and the initiation of study medication
8. Patient report of dyspnea at rest or upon minimal exertion during screening at least one hour after administration of IV loop diuretic

Exclusion Criteria:

1. Women who are pregnant or breast-feeding
2. Clinical presentation:

   1. Suspected ACS based on clinical judgment
   2. Coronary revascularization in the 3 months prior to screening or planned during current admission.
   3. Temperature >38.5oC
   4. Clinically significant anemia
   5. Serum sodium >145 mEq/L (145 mmol/L)
   6. Current or planned ultrafiltration, paracentesis, hemofiltration or dialysis at time of screening
   7. Any mechanical ventilation
   8. CPAP/BiPAP discontinued less than 1 hour prior to randomization
   9. History of LVAD or IABP within the last year
   10. Intravenous radiographic contrast agent within 72 hours prior to screening or presence of acute contrast induced nephropathy at the time of screening
   11. Presence of clinically significant arrhythmia
   12. Uncertainty of ability to complete follow up
3. Medications:

   1. nitroprusside or nesiritide
   2. Intravenous nitrates
   3. use of inotropes
   4. Use of ARBs within 7 days of prior to randomization
   5. Use of any investigational medication within 30 days
   6. clinically significant hypersensitivity or allergy to, or intolerance of, angiotensin receptor blockers
4. Medical history:

   1. Major surgery within 8 weeks prior to screening
   2. Stroke within 3 months prior to screening
   3. eGFR (sMDRD) <20 mL/min/1.73m2 or >75 mL/min/1.73m2 between presentation and randomization
   4. Post cardiac or renal transplant
   5. Listed for renal transplant or cardiac transplant with anticipated transplant time to transplant < 6 months
   6. History of severe left ventricular outlet obstruction (either valvular or sub-valvular), severe mitral valve stenosis or severe aortic regurgitation
   7. Cardiac valvular abnormality that requires surgical correction
   8. Complex congenital heart disease
   9. Hypertrophic or restrictive cardiomyopathy
   10. significant pulmonary or hepatic disease that could interfere with the evaluation of safety or efficacy of TRV027
   11. life expectancy of less than 6 months

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
composite z score | 30 days
  The primary clinical endpoint is a of the following outcomes: (1) time from randomization to death through day 30, (2) time from randomization to heart failure re-hospitalization through day 30, (3) time from randomization to worsening heart failure through day 5, (4) change in dyspnea VAS score (calculated area under the curve) from baseline through day 5, and (5) length of initial hospital stay (in days) from randomization. The component outcomes will be combined by deriving an average Z for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: David Soergel, MD, Study Director — Trevena Inc.
Locations (62):
- United States (4):
  - Wayne State University, Detroit, Michigan
  - University of Cincinnati, Cincinnati, Ohio
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Michael E Debakey VA Medical Center, Houston, Texas
- Argentina (11):
  - Research Site, Buenos Aires
  - Research Site, Coronel Suárez
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Morón
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Martín
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Bulgaria (7):
  - Research Site, Dimitrovgrad
  - Research Site, Kazanlak
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Smolyan
  - Research Sites, Sofia
  - Research Site, Sofia
- Canada (2):
  - Research Site, Edmonton, Alberta
  - Research Site, Ottawa, Ontario
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- Germany (3):
  - Research Site, Berlin
  - Research Site, Dortmund
  - Research Site, Greifswald
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Kaposvár
  - Research Site, Pécs
- Israel (8):
  - Research Site, Afula
  - Research Site, Ashkelon
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Nazareth
  - Research Site, Safed
- Poland (9):
  - Research Site, Bad Nauheim
  - Research Site, Bialystok
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Krakow
  - Research Site, Kłodzko
  - Research Site, Lublin
  - Research Site, Ruda Śląska
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (5):
  - Research Site, Baia Mare
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Târgu Mureş
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Kocise
  - Research Site, Martin